CLINICAL TRIAL: NCT07392411
Title: Study on Artificial Intelligence-Based Facial and Speech-Related Patterns in Parkinson's Disease and Their Digital Biomarkers
Status: Recruiting | Type: Observational
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 7232048
Record Dates: First submitted 2026-01-30; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Parkinson's Disease; Progressive Supranuclear Palsy(PSP); Multiple System Atrophy; Healthy Control
MeSH Terms: conditions — Parkinson Disease; Supranuclear Palsy, Progressive; Multiple System Atrophy | interventions — Videotape Recording

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Parkinson's disease (PD) group: Participants meeting the 2015 MDS clinical diagnostic criteria for PD, aged 18-75. Includes both early (Hoehn-Yahr stage 1-2.5) and advanced (Hoehn-Yahr stage 2.5-5) patients. All participants provide informed consent for facial video and speech audio data collection. Exclusion criteria: history of stroke, head trauma, hydrocephalus, brain tumors, intracranial surgery, metal implants, pacemakers, severe dyskinesia, or MMSE score ≤ 24.
  Interventions: Other: video recording
- Multiple System Atrophy (MSA) Group: Participants diagnosed with MSA-P according to the 2017 Chinese expert consensus diagnostic criteria, aged 18-75. For unified motor assessment, MDS-UPDRS I-IV and Hoehn-Yahr staging are used. All provide informed consent for data collection. Exclusion criteria: history of stroke, head trauma, hydrocephalus, brain tumors, intracranial surgery, metal implants, pacemakers, or MMSE score ≤ 24.
  Interventions: Other: video recording
- Progressive Supranuclear Palsy (PSP) Group: Participants diagnosed with PSP according to the 2016 Chinese clinical diagnostic criteria, aged 18-75. For unified motor assessment, MDS-UPDRS I-IV and Hoehn-Yahr staging are used. All provide informed consent for data collection. Exclusion criteria: history of stroke, head trauma, hydrocephalus, brain tumors, intracranial surgery, metal implants, pacemakers, or MMSE score ≤ 24.
  Interventions: Other: video recording
- Healthy Control Group: Age- and sex-matched healthy volunteers with no neurological diseases. MMSE score ≥ 24. All participants provide informed consent and undergo the same standardized facial video and speech audio recording tasks as the patient groups. Exclusion criteria: history of any neurological or psychiatric disorders.
  Interventions: Other: video recording

INTERVENTIONS:
Other: video recording — The patient's facial expressions and speech characteristics were recorded via video for assessment purposes.

SUMMARY:
This research employs AI to analyze facial expressions and speech patterns, aiming to develop new digital tools for diagnosing and differentiating Parkinson's disease and similar disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for Parkinson's Disease (PD) Group: (1) Diagnostic Criteria: Meet the diagnostic criteria for Parkinson's disease established by the Movement Disorder Society (MDS) in 2015. (2) Age Range: 18-75 years old. (3) Disease Severity: Early-stage PD: Hoehn-Yahr score ≤ 2.5 points. Mid-to-late-stage PD: Hoehn-Yahr score 2.5-5 points. (4) Consent for Data Collection: Willing to undergo facial expression video and speech audio recording. (5) Informed Consent: Signed informed consent form.
2. Inclusion Criteria for Parkinson's Plus Syndromes (MSA-P, PSP) Group: (1) Age Range: 18-75 years old. (2) Diagnostic Criteria: MSA patients must meet the diagnostic criteria established by the [Chinese Expert Consensus on the Diagnosis of Multiple System Atrophy, 2017]. PSP patients must meet the diagnostic criteria established by the [Chinese Clinical Diagnostic Criteria for Progressive Supranuclear Palsy, 2016 Edition]. (3) Consent for Data Collection: Willing to undergo facial expression video and speech audio recording. (4) Informed Consent: Signed informed consent form.

Exclusion Criteria:

1. History of cerebrovascular disease, head trauma, hydrocephalus, brain tumors, or intracranial surgery.
2. Presence of metal implants, cardiac pacemakers, or other metallic foreign bodies (applies to PD patients).
3. Severe dyskinesia in PD patients that would compromise cooperation with video/audio recording.
4. Mini-Mental State Examination (MMSE) score ≤ 24 points.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In this study, participants were recruited from a single center in China. They were enrolled through outpatient assessment and screening.
Sampling Method: Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic Accuracy of the AI Model in Assessing [ Disease/Condition ] Severity | Baseline
  The effectiveness of the model was demonstrated through a comparison between model-predicted scores and human expert ratings.

CONTACTS AND LOCATIONS:
Locations (1):
- 首都医科大学附属北京天坛医院, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data will not be publicly available, but can be shared with collaborators under specific agreements.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code